CLINICAL TRIAL: NCT07060742
Title: Feasibility of Exergame-based Cognitive-motor Training in Older Psychotic Inpatients: a Randomized Controlled Trial
Brief Title: Study on the Use of Exergames to Support Older Adults With Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tobias Melcher (Network)
Responsible Party: Sponsor-Investigator, Tobias Melcher, Dr. Dipl.-Psych. Tobias Melcher, Principal Investigator of the study, University Psychiatric Clinics Basel
Organization: University Psychiatric Clinics Basel (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dividat-Psychosen25
Record Dates: First submitted 2025-06-16; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Psychosis; Exergaming; Elderly
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dividat Senso (Exergame-Based Motor-Cognitive Training) (Experimental): Participants in this group will receive the standard psychiatric inpatient care at the Psychiatric University Hospital Basel. In addition, they will engage in technology-based motor-cognitive training using the Dividat Senso device. This system involves interactive exergames that require participants to perform body movements such as stepping and shifting weight in response to multisensory stimuli (visual, auditory, and somatosensory). The games are designed to simultaneously stimulate physical functions (balance, coordination) and cognitive functions (attention, executive function, memory). Training sessions will be conducted three times a week for four weeks, with each session lasting approximately 20 minutes, totaling 12 sessions.
  Interventions: Device: Dividat Senso
- OTAGO Falls-Prevention Program (Traditional Strength and Balance Exercises) (Active Comparator): Participants in the control group will also receive the standard psychiatric inpatient care. Additionally, they will participate in conventional physical exercises focusing on strength and balance, based on the Otago falls prevention program. These exercises are designed to improve physical stability and reduce fall risk. Like the intervention group, participants will train three times a week for four weeks, with each session lasting about 20 minutes, totaling 12 sessions.
  Interventions: Other: OTAGO Falls-prevention program

INTERVENTIONS:
Device: Dividat Senso — Participants in the intervention group will receive cognitive-motor training using the Dividat Senso exergame platform, which records body movements and adapts game difficulty in real time. The training targets cognitive and physical functions through interactive games involving steps and weight shifts. It follows a progressive structure, with difficulty increasing over time, and can be personalized by investigators using the Dividat Manager.
  Arms: Dividat Senso (Exergame-Based Motor-Cognitive Training)
Other: OTAGO Falls-prevention program — The OTAGO Falls Prevention Program is an evidence-based exercise program designed to reduce falls in older adults. It includes strength and balance training exercises performed at home under the guidance of a physiotherapist. The program aims to improve muscle strength, balance, and mobility, helping to prevent falls and maintain independence.
  Arms: OTAGO Falls-Prevention Program (Traditional Strength and Balance Exercises)

SUMMARY:
This study aims to explore a new, engaging approach to support older adults with psychosis-an umbrella term that includes conditions such as schizophrenia, late-onset schizophrenia, and psychotic symptoms resulting from other medical or psychiatric conditions like dementia, delirium, mood disorders, or delusional disorder. As the aging population grows, a rising number of older adults are living with schizophrenia and related disorders, facing not only psychiatric symptoms like hallucinations and delusions but also cognitive impairments, reduced mobility, social isolation, and physical decline. These combined challenges significantly affect daily functioning and quality of life. At present, there are no psychosis treatment guidelines specifically tailored for people aged 60 and above, though general principles from younger populations can be adapted. Evidence suggests that integrating physical and cognitive rehabilitation into standard psychiatric care may enhance treatment outcomes for this age group. One promising method is the use of "exergames"-interactive video games that combine physical movement with cognitive challenges. These games typically require users to perform body movements such as stepping or shifting weight in response to visual and auditory cues, thereby training functions like attention, memory, balance, coordination, and executive function. Exergames offer a playful and stimulating alternative to conventional exercises and are often better accepted by older patients because of their engaging and motivating nature. Previous studies have shown that older adults with schizophrenia not only tolerate these games well but may also experience improvements in mood, cognitive function, and physical activity levels. However, past research has been limited by small sample sizes, lack of control groups, and short intervention periods. This current study, conducted at the Psychiatric University Hospital in Basel, Switzerland, seeks to examine the feasibility and benefits of using an exergame system called Dividat Senso in a more structured and controlled setting. After being screened for eligibility, participants will be randomly assigned to one of two groups. The intervention group will receive usual psychiatric inpatient care, extended with exergame-based motor-cognitive training using the Dividat Senso platform. This device requires full-body interaction, targeting both cognitive functions (such as attention, memory, and executive skills) and physical abilities (such as balance and coordination). The control group will also receive usual care, but instead of exergames, they will participate in traditional strength and balance exercises taken from the Otago falls prevention program. Both groups will train three times a week for four weeks, with each session lasting approximately 20 minutes-totaling 12 sessions. All participants will complete assessments before the intervention begins (T1) and again after four weeks (T2), to measure changes in physical activity, mental well-being, and cognitive performance. By using a structured program and comparing two active interventions, this study aims to generate more robust and generalizable findings on how technology-based, body-and-brain training can support the mental and physical health of older adults with psychosis. If proven feasible and effective, exergame-based rehabilitation could become a valuable and enjoyable addition to psychiatric treatment programs for elderly patients.

DETAILED DESCRIPTION:
Elderly patients with psychosis can be categorized into three groups: those with a history of schizophrenia, those with a new diagnosis of schizophrenia (late-onset), and those experiencing hallucinations or delusions due to other conditions such as dementia, delirium, delusional disorder, mood disorders, or paranoid personality disorders. The elderly population with schizophrenia represents a growing segment of older adults, with an estimated prevalence of 4-6% among people over 65 years old and around 10% among those over 85. Core features associated with psychosis include hallucinations, which are perceptions without external stimuli, and delusions, which are fixed false beliefs maintained despite evidence to the contrary. Other symptoms linked to psychosis include thought interference, thought disorder, apathy, social withdrawal, and blunted affect. Currently, there are no specific guidelines for managing primary psychotic disorders in adults aged 60 and older, but some general principles can be adapted from guidelines for other age groups. Existing recommendations for adults under 60 emphasize addressing not only psychiatric symptoms but also other health factors that affect overall well-being. Given the significant impact of cognitive and physical impairments, social isolation, and sensory deficits on symptoms in older adults, an integrated approach addressing both mental and physical health could improve treatment outcomes in this population. Research has shown that greater severity of schizophrenia symptoms and neurocognitive impairments are associated with reduced levels of physical activity, and that effective physical activity interventions should include components that enhance cognition and reduce psychiatric symptoms. One specific form of physical activity is exergaming, which combines physical exercise with cognitive stimulation through gameplay. Exergames involve multisensory stimuli, including auditory, visual, and somatosensory modalities, requiring engagement of various cognitive functions such as executive functions, visual and verbal memory, attention, and other multidimensional cognitive processes. Exergames offer several advantages over conventional exercise in enhancing cognitive functions by integrating cognitive demands into physical tasks. Furthermore, exergames promote better long-term adherence to exercise due to their gamified and motivational nature. Previous studies suggest that video game-based physical activity programs have higher acceptability and adherence rates among older adults with schizophrenia. Similar results were observed in chronic psychiatric inpatient populations, where full-body interaction during computerized cognitive training led to cognitive improvements and reduced depressive symptoms. Additionally, video game-based physical activity programs have increased the frequency of self-reported physical activity among older adults with schizophrenia. Meta-analytical evidence suggests that virtual reality exergames may positively influence cognition and depression in older populations. However, current evidence is limited by small sample sizes, low participant heterogeneity, inadequate training duration and frequency, and lack of control groups. To obtain generalizable findings on the feasibility and effects of exergame-based motor-cognitive training in inpatient settings for older patients with psychosis, future research should include frequent, structured training sessions, heterogeneous samples, and control groups. Technological advancements over recent decades have increased the availability of digitalized motor-cognitive training options. One such option is the use of a "step plate" for exergame training, such as the Dividat Senso. These exergames specifically target cognitive functions essential for daily living, including executive functions, attention, as well as physical abilities like balance and coordination. The games are played through body movements and weight shifting. To examine the feasibility and effects of exergame-based motor-cognitive training in older psychiatric inpatients, we plan to use the Dividat Senso device. After eligibility screening, participants undergo baseline assessment (T1) and are randomly assigned to one of two groups. The intervention group receives conventional treatment at the psychiatric hospital extended by technology-based motor-cognitive training using Dividat Senso. The control group receives conventional treatment plus strength and balance exercises from the Otago falls-prevention program. The intervention lasts four weeks, with participants requested to engage in short training sessions three times per week for 20 minutes each, totaling 12 sessions. After the intervention period, all participants undergo a post-intervention assessment (T2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed psychotic disorders
* Able to provide a signed informed consent
* Age ≥ 55 years
* MoCA ≥ 20
* Physically able to stand for at least 3 minutes without external support (self-report)

Exclusion Criteria:

* Insufficient knowledge of the German language to understand the instructions, the games, and the assessments
* Mobility, cognitive, sensory and/or psychiatric limitations or comorbidities that impair the ability to play the exergames and/or conduct the pre-/post assessments

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the exergame-based motor-cognitive training: adherence | Throughout the 4-week intervention period.
  The adherence protocol measures the percentage of training sessions attended by participants relative to the number of planned sessions. It reflects how consistently participants follow the prescribed training schedule. Adherence is calculated by dividing the attended sessions by the planned sessions and expressing the result as a percentage. High adherence rates suggest that the intervention is feasible for older psychotic inpatients.
Feasibility of the exergame-based motor-cognitive training: attrition | Time Frame: Throughout the 4-week intervention period
  Attrition: Drop-Out Rates. This refers to the percentage of participants who discontinue or leave the study before its completion. Drop-out rates are calculated by dividing the number of participants who withdraw by the total number initially enrolled, usually expressed as a percentage. High dropout rates may indicate issues with the intervention's feasibility.
Feasibility of the exergame-based motor-cognitive training: safety | Time Frame: Throughout the 4-week intervention period
  Safety, measured through the reporting of adverse events, assesses the occurrence and nature of any negative or unintended effects experienced by participants during the study. These events are systematically recorded, including their type, severity, timing, and potential relation to the intervention. No adverse events indicate that the intervention is safe and feasible.

SECONDARY OUTCOMES:
Cognitive function: inhibitory control | Throughout the 4-week intervention period
  Stroop Color and Word Test (Senso-based):
  This test measures inhibitory control. Participants are shown words that name colors (e.g., "blue", "red") printed in incongruent ink colors (e.g., the word "blue" printed in red ink). They must name the color of the ink, not read the word, requiring them to suppress the automatic reading response. Reaction time (in milliseconds) and accuracy are recorded. Lower reaction times and fewer errors indicate better executive functioning.
Cognitive function: processing speed | Time Frame: Throughout the 4-week intervention period
  Reaction Time Test (RTT, Senso-based):
  This test measures basic processing speed. Participants are presented with simple visual stimuli on a screen (e.g., a light or symbol) and must respond as quickly as possible by pressing a button or stepping onto a platform. The test records reaction time in milliseconds and the number of errors (e.g., missed or premature responses). Shorter reaction times and fewer errors indicate better cognitive and motor responsiveness.
Cognitive function: selective attention | Time Frame: Throughout the 4-week intervention period
  Arrow Test (Senso-based):
  This test assesses inhibitory control. It consists of two phases:
  * In the first phase, participants stand on a central platform and must step toward the side where an arrow appears on the screen, reacting as quickly as possible.
  * In the second phase, participants must step in the direction the arrow points, regardless of its position on the screen (e.g., an arrow may appear on the left but point to the right), requiring greater cognitive control to inhibit automatic responses.
  Reaction time (ms) and number of errors are recorded. Lower reaction times and fewer errors indicate better performance.
Cognitive function: inhibitory control | Time Frame: Throughout the 4-week intervention period
  The Go-NoGo Test (Senso-based) primarily measures inhibitory control. Participants focus on a central gray dot while an "x" or "+" appears to the left or right. When an "x" appears, they must quickly step toward its location; when a "+" appears, they must withhold any response. Reaction time (in milliseconds) and accuracy-both correct responses to "x" and successful inhibitions to "+"-are recorded. Lower reaction times and higher accuracy indicate better cognitive control and response inhibition.
Motor function: mobility | Time Frame: Throughout the 4-week intervention period
  The Timed Up and Go Test (TUG) measures functional mobility. Participants start seated in a chair, then stand up, walk a short distance (usually 3 meters), turn around, walk back, and sit down again. The time taken to complete this sequence is recorded in seconds. The test is performed under both single-task (just walking) and dual-task conditions (walking while performing a cognitive or motor task). Shorter times indicate better mobility, balance, and ability to perform everyday movements safely and efficiently.
Motor function: gait speed | Time Frame: Throughout the 4-week intervention period
  The 10-Meter Walk Test measures gait speed. Participants are asked to walk a 10-meter distance twice: once at their normal, comfortable pace, and once at an accelerated, faster pace. The time taken to complete each walk is recorded in seconds, and gait speed is calculated by dividing distance by time. Higher gait speeds indicate better walking performance, mobility, and functional capacity.
Motor function: balance | Time Frame: Throughout the 4-week intervention period
  The Coordinated Stability Test (Senso-based) measures balance coordination. Participants stand still and adjust their body by bending or rotating-without moving their feet-to keep a cursor or marker within a designated track displayed on the screen. The test records metrics such as completeness and stability (where higher values indicate better control), as well as path length, duration, and reverse movements (where lower values indicate better performance). This assesses the ability to maintain balance and make fine motor adjustments to remain stable.
Motor function: physical activity | Time Frame: Throughout the 4-week intervention period
  The accelerometers ActiGraph GT3X+ and Axivity AX3 measure physical activity levels by continuously recording tri-axial acceleration data over a 48-hour period. Worn on the body, these devices capture movement intensity and frequency. The raw acceleration data are processed and classified into different activity intensity categories-such as sedentary, light, moderate, and vigorous-based on predefined thresholds. Higher activity counts indicate more intense or frequent movement, while lower counts reflect periods of inactivity or sedentary behavior. This allows objective assessment of overall physical activity patterns and sedentary time.
Psychotic symptoms: patient's response to treatment | Time Frame: Throughout the 4-week intervention period
  The Clinical Global Impression of Change (CGI) measures overall symptom severity and the patient's response to treatment, as rated by a clinician. Using standardized scales, the clinician assesses how much the patient's condition has improved or worsened compared to baseline. Lower scores indicate fewer symptoms and better treatment response, while higher scores reflect more severe symptoms or less improvement. This tool provides a quick, global evaluation of clinical status and treatment effectiveness. The Severity of Illness scale includes: Not assessable; Not ill at all; Borderline psychiatric case; Mildly ill; Moderately ill; Markedly ill; Severely ill; Extremely severely ill.The Global Improvement scale includes: Not assessable; Very much improved; Much improved; Slightly improved; No change; Slightly worse; Much worse; Very much worse
Psychotic symptoms: severity of psychotic symptoms | Time Frame: Throughout the 4-week intervention period
  The Positive and Negative Syndrome Scale (PANSS) measures the severity of psychotic symptoms across three domains: positive symptoms (e.g., hallucinations, delusions), negative symptoms (e.g., social withdrawal, lack of motivation), and general psychopathology (e.g., anxiety, depression). A clinician rates each of the 30 items on a standardized scale from 1 to 7, where 1 = Absent, 2 = Minimal, 3 = Mild, 4 = Moderate, 5 = Moderately severe, 6 = Severe, and 7 = Extreme. Scores are summed to produce total and subscale scores. Higher scores indicate more severe symptoms, while lower scores reflect milder symptom severity. The PANSS is widely used to assess and monitor the clinical status of patients with psychotic disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Melcher, Dr. Dripl.Psych., Study Director — Universitäre Psychiatrischen Kliniken (UPK) Basel
Locations (1):
- Universitäre Psychiatrischen Kliniken (UPK) Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yen HY, Chiu HL. Virtual Reality Exergames for Improving Older Adults' Cognition and Depression: A Systematic Review and Meta-Analysis of Randomized Control Trials. J Am Med Dir Assoc. 2021 May;22(5):995-1002. doi: 10.1016/j.jamda.2021.03.009. Epub 2021 Apr 2. PMID 33812843
- [Background] Maillot P, Perrot A, Hartley A. Effects of interactive physical-activity video-game training on physical and cognitive function in older adults. Psychol Aging. 2012 Sep;27(3):589-600. doi: 10.1037/a0026268. Epub 2011 Nov 28. PMID 22122605
- [Background] Leutwyler H, Hubbard EM, Jeste DV, Vinogradov S. "We're not just sitting on the periphery": a staff perspective of physical activity in older adults with schizophrenia. Gerontologist. 2013 Jun;53(3):474-83. doi: 10.1093/geront/gns092. Epub 2012 Aug 30. PMID 22936534
- [Background] Leutwyler H, Hubbard EM, Jeste DV, Miller B, Vinogradov S. Associations of schizophrenia symptoms and neurocognition with physical activity in older adults with schizophrenia. Biol Res Nurs. 2014 Jan;16(1):23-30. doi: 10.1177/1099800413500845. Epub 2013 Sep 19. PMID 24057223
- [Background] Leutwyler H, Hubbard EM, Dowling GA. Adherence to a Videogame-Based Physical Activity Program for Older Adults with Schizophrenia. Games Health J. 2014 Aug;3(4):227-33. doi: 10.1089/g4h.2014.0006. Epub 2014 May 28. PMID 26192371
- [Background] Leutwyler H, Hubbard E, Cooper B, Dowling G. The Impact of a Videogame-Based Pilot Physical Activity Program in Older Adults with Schizophrenia on Subjectively and Objectively Measured Physical Activity. Front Psychiatry. 2015 Dec 21;6:180. doi: 10.3389/fpsyt.2015.00180. eCollection 2015. PMID 26733891
- [Background] Camara J, Ferreira L, Faria AL, Vilar M, Bermudez I Badia S. Feasibility, Acceptability, and Preliminary Impact of Full-Body Interaction on Computerized Cognitive Training Based on Instrumental Activities of Daily Living: A Pilot Randomized Controlled Trial with Chronic Psychiatric Inpatients. Games Health J. 2022 Oct 11. doi: 10.1089/g4h.2021.0228. Online ahead of print. PMID 36251861
- See also: The Dividat Senso is a scientifically validated exergame platform that combines cognitive and physical training through interactive step-based games, enhancing balance, coordination, and mental function in older adults and clinical populations. — https://dividat.com/senso